CLINICAL TRIAL: NCT01904227
Title: A Randomized Controlled Study of the Efficacy of an Intensified, Inpatient Adaptation of Dialectical Behavior Therapy (DBT) for a Population of Borderline Patients (Young Adults/Adults: 18 - 40), Compared With Standard Outpatient DBT.
Brief Title: Intensified, Inpatient Adaptation of Dialectical Behavior Therapy (DBT)
Acronym: REDBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GGZ Rivierduinen (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rivierduinen 2012
Record Dates: First submitted 2013-07-11; First posted 2013-07-22 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Dialectical Behavior Therapy
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inpatient Adaptation of DBT (Experimental): Patients are in treatment 5 days a week, during 12 weeks. Staff is only present in daytime. During the weekends the patients stay at home.
  The therapy consists of DBT skills training (Linehan, 1996), individual psychotherapy (Linehan, 2002), crisis consultation if needed, and weekly meetings of the consultation team for all trainers and therapists for one hour. Staff also receives supervision twice-weekly.
  Patients also receive daily mindfulness classes, 2 hours of drama therapy, psycho educational classes about sexuality, substance abuse and medication, and the possibility to get help in applying principles of validation and behavioral analysis skills.
  Interventions: Behavioral: Inpatient Adaptation of DBT
- Outpatient DBT (Active Comparator): Control condition: Standard outpatient DBT
  Interventions: Behavioral: standard outpatient DBT

INTERVENTIONS:
Behavioral: standard outpatient DBT — Patients receive 12 months of outpatient treatment as specified in the DBT manual (Linehan, 2002) in one of the participating regional psychiatric centers of Rivierduinen. The treatment is according to protocol and combines weekly individual cognitive-behavioral psychotherapy sessions with the primary therapist, weekly skills- training groups, if needed consultation and weekly consultation meetings for trainers and therapists.
  Arms: Outpatient DBT
Behavioral: Inpatient Adaptation of DBT — The intervention to be studied, inpatient DBT, consists of an inpatient program of 12 weeks. The department provides accommodation for 9 patients. Patients are admitted 5 days a week at the department Oost, part of the Jelgersma centre for Personality Disorders. Staff is only present in daytime. During the weekends the patients stay at home.
  The therapy consists of DBT skills training (Linehan, 1996), individual psychotherapy (Linehan, 2002), crisis consultation if needed, and weekly meetings of the consultation team for all trainers and therapists for one hour. Staff also receives supervision twice-weekly.
  Arms: Inpatient Adaptation of DBT

SUMMARY:
An randomized clinical trial to investigate whether among adult borderline patients (18 - 40 year), intensified inpatient short term (12 weeks) inpatient Dialectical Behavior Therapy (DBT) is more effective in declining the proportion of patients that show suicidal/self-harming behavior in the first 3 months of treatment, compared to standard outpatient DBT, and whether this difference between the groups is sustained at 6 and 12 months.

DETAILED DESCRIPTION:
Objective: Goal is to evaluate the (cost-)effectiveness of a short term intensive DBT treatment program (12 weeks) versus outpatient DBT, in terms of reduction of suicidal and/or self-harming behavior, and of general BPD symptomatology severity.

Study design: A randomized trial, analyzed by a intention-to-treat (ITT) approach, with two parallel groups: a) intensified adapted DBT program (12 weeks inpatient program, plus six months standard outpatient DBT, n=36); b) standard outpatient DBT for 12 months (n=36).

Study population: All borderline patients (18-40 years), who will be admitted from January 2013 till June 2014 for treatment in the Jelgersma Treatment Centre, or the outpatient DBT programs of Rivierduinen, who: (1) receive a diagnosis of BPD, (2) have shown suicidal and/or self-harming behavior in the year preceding the admission/ start of DBT treatment, including the last month preceding baseline measurement, and (3) show a severe level of borderline symptomatology (> 24 on the BPDSI).

Intervention:

All patients receive DBT according to the basic DBT treatment protocol. Treatment integrity is established by supervision in both groups.

Outcome measures Main study parameter is the number of suicide attempts/self-harming acts (the Life Time Parasuicide Count and the Parasuicide Scale of the Borderline Personality Severity Index). Second study parameter is the severity of borderline symptomatology (BPDSI). Quality of life as measured on the SF-36, and the EQ-5D and psychopathological symptoms (BSI) will also be taken into account. The cost-effectiveness of the inpatient program compared to the outpatient program will be examined (TiC-P).

Sample size. The researchers expect that after 12 weeks of treatment, 20% of the patients of the intervention group still show suicidal and/or self-harming behavior compared to 60% of the patients in the control condition, and that this difference sustains after 24 weeks and will be gradually reduced between 24 and 52 weeks by the additional reduction in suicidal and/or self-harming behavior in the control group. To be able to detect a difference of 40% after 12 weeks, with a power of 0.80 and α = 0.05, 36 patients per experimental condition are required. The researchers expect to recruit about 150 patients, which guarantees enough power, even with a 20% drop out rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in the period of January 2013 until January 2014
* patients who fulfill the Diagnostic and Statistical Manual-IV Text Revision criteria for BPD,
* patients who have shown suicidal and/or self-harming behavior in the year preceding the admission/ start of DBT treatment, including the last month preceding baseline measurement,
* patients who show a severe level of borderline symptomatology ( > 24 on the BPDSI),
* patients who are in sufficient command of the Dutch language

Exclusion Criteria::

* Intelligence Quotient < 80,
* a chronic psychotic condition,
* bipolar disorder,
* hard drug abuse that requires inpatient detoxification,
* forced treatment framework,
* DBT in the year preceding intake.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
assessing change in number of suicide attempts/self-harming acts | baseline, 0, 12, 24 and 52 weeks after the start of the inpatient treatment
  The Lifetime Parasuicide Count (LPC: Comtois & Linehan, 1999), obtains information about the frequency and subsequent medical treatment of self-mutilating behaviors (e.g. cutting, burning and pricking). Duration of the interview depends on how frequent and how much self-destructive behavior has been shown. Patients report that they feel that their problems are taken seriously because of the interview.
  The Borderline Personality Disorder Severity Index (BPDSI: (Giessen-Bloo et al., 2010) is a semi-structured interview assessing the frequency of borderline symptoms in the previous 3-month period. The BPDSI consists of nine sections, one for each of the Diagnostic and Statistical Manual-IV criteria for borderline personality disorder. The parasuicide section includes three items reflecting distinct suicidal behaviors (suicide threats, preparations for suicide attempts, and actual suicide attempts).

SECONDARY OUTCOMES:
assessing change in the severity of borderline symptomatology | at baseline, 0, 12, 24 and 52 weeks after the start of the inpatient treatment
  The Borderline Personality Disorder Severity Index (BPDSI: (Giessen-Bloo et al., 2010) is a semi-structured interview assessing the frequency of borderline symptoms in the previous 3-month period. The BPDSI consists of nine sections, one for each of the criteria for borderline personality disorder from the Diagnostic and Statistical Manual-IV.The parasuicide and impulsivity sections have shown reasonable internal consistencies (0.69 and 0.67, respectively), excellent interrater reliability (0.95 and 0.97, respectively) and good concurrent validity ( Arntz et al., 2003). Three month test-retest reliability for the total BPDSI score was 0.77. Patients have reported that they feel acknowledged by the BPDSI for their problems (van den Bosch, 2005).

OTHER OUTCOMES:
assessing change in level of Quality of life | baseline, 0, 12, 24 and 52 weeks after the start of the inpatient treatment
  The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being: Physical Functioning (10 items), Role-Physical (4 items), Bodily Pain (2 items), General Health (5 items), Vitality (4 items), Social Functioning (2 items), Role-Emotional (3 items) and Mental Health (5 items) as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.
  The EuroQol 5 Dimensions descriptive system (EQ-5D) consists of five dimensions (Mobility, Self Care, Usual Activities, Pain/Discomfort and Anxiety/Depression) with three levels each (no problems, some problems and extreme problems), thus defining 243 (35) distinct health states.
assessing the cost-effectiveness of the inpatient program compared to the outpatient program | baseline and 52 weeks after the start of the inpatient treatment
  The 'Trimbos and institute for Medical Technology Assessment questionnaire on Costs associated with Psychiatric illness' (TiC-P: Hakkaart- van Roijen, 2010) is a validated tool commonly applied in economic evaluations of treatments in mental health care. The TiC-p consists of two parts. The first part measures direct medical costs. The second part estimates the productivity costs. The number of hospital days and/or outpatient contacts for treatment will also be collected directly from the participating centres. Reference unit prices of health care services will be applied (Hakkaart et al, 2010).
  The second part of the TiC-P includes a short form of the Health and Labor questionnaire (HLQ) for collecting data on productivity losses (van Roijen et al., 1996).
assessing change in level of psychopathological symptoms | baseline, 0, 12, 24 and 52 weeks after the start of the inpatient treatment
  The Brief Symptomatology Inventory (BSI; Derogatis & Melisaratos, 1983) includes 49 items grouped into nine scales that encompass nine primary dimensions of psychopathological symptoms: psychoticism, somatization, depression, hostility, phobic anxiety, obsessive-compulsivity, anxiety (panic), paranoid ideation, and nervous tension. As to reliability, Derogatis and Melisaratos (1983) presented appropriate coefficients of internal consistency of the BSI ranging from 0.71 to 0.85 and test-retest reliability coefficients ranging from 0.68 to 0.91. Other studies have reported similar estimates (e. g., Boulett & Boss, 1991; Hayes, 1997). As to validity, Derogatis and Melisaratos (1983) provided evidence for a good construct validity of the BSI.

CONTACTS AND LOCATIONS:
Overall Officials: Louisa M van den Bosch, PhD, Principal Investigator — GGZ Rivierduinen
Locations (1):
- LMC van den Bosch, Oegstgeest, Netherlands

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Sinnaeve R, van den Bosch LMC, Hakkaart-van Roijen L, Vansteelandt K. Effectiveness of step-down versus outpatient dialectical behaviour therapy for patients with severe levels of borderline personality disorder: a pragmatic randomized controlled trial. Borderline Personal Disord Emot Dysregul. 2018 Jul 10;5:12. doi: 10.1186/s40479-018-0089-5. eCollection 2018. PMID 30002832